CLINICAL TRIAL: NCT02352896
Title: Long-Term Safety and Efficacy Evaluation of Vatiquinone (EPI-743) in Children With Leigh Syndrome
Brief Title: Long-Term Safety and Efficacy Evaluation of EPI-743 in Children With Leigh Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI743-13-023
Record Dates: First submitted 2014-08-21; First posted 2015-02-02 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Leigh Syndrome
Keywords: Leigh syndrome; Mitochondrial disorders; EPI743; Vincerinone
MeSH Terms: conditions — Leigh Disease; Mitochondrial Diseases | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-743 (Experimental): Participants will receive EPI-743 at a dose of 15 milligrams/kilogram (mg/kg) up to a total 200 mg 3 times daily (TID) orally with meal or by using nasogastric (NG) or gastrostomy feeding tubes with liquid food for at least 36 months.
  Interventions: Drug: EPI-743

INTERVENTIONS:
Drug: EPI-743 — EPI-743 100 milligrams/milliliter (mg/mL) oral solution will be administered per dose and schedule specified in the arm.
  Other Names: Vincerinone, Vatiquinone

SUMMARY:
EPI-743 in Leigh syndrome participants that participated in previous EPI743-12-002 (NCT01721733) study.

DETAILED DESCRIPTION:
To monitor the long-term safety and neurodevelopmental effects of EPI-743 on children who complete the EPI743-12-002 placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Leigh syndrome with genetic confirmation
2. Completion of EPI743-12-002 protocol and initiation of treatment within 14 days of Month 12 visit in EPI743-12-002 study
3. Participant or participant's guardian able to consent and comply with protocol requirements
4. Continued abstention from supplements excluded in EPI743-12-002 study
5. Botox® is allowed if approved by the sponsor

Exclusion Criteria:

1. Allergy to EPI-743 or sesame oil
2. Allergy to vitamin E
3. Clinical history of bleeding or abnormal baseline prothrombin time (PT)/partial thromboplastin time (PTT)
4. Hepatic insufficiency with liver function tests (LFTs) greater than two times upper limit of normal
5. Renal insufficiency requiring dialysis
6. End-stage cardiac failure
7. Fat malabsorption syndromes precluding drug absorption
8. Use of anticoagulant medications
9. Participation in other clinical research studies/taking other experimental agents
10. Participation in elective procedures that required sedation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Disease Severity as Measured by Newcastle Pediatric Mitochondrial Disease Scale (NPMDS) Sections 1-3 Score | Baseline up to Month 36
  NPMDS is a validated scale to assess the mitochondrial disease progression.
Number of Participants With Dose-Limiting Serious Adverse Events (SAEs) | Baseline up to Month 36

SECONDARY OUTCOMES:
Bayley Scales of Infant Development-III Score (Participants Age 0-3) | Baseline up to Month 24
  Effect of EPI-743 on neurodevelopment will be measured by Bayley Scales of Infant Development-III score.
Wechsler Scale of Intelligence and Movement Assessment Battery Score for Children (Participants Age 4-18) | Baseline up to Month 24
  Effect of EPI-743 on neuromuscular function will be assessed by Wechsler Scale of Intelligence and Movement Assessment Battery score.
Barry-Albright Dystonia Scale Score | Baseline up to Month 24
  Neuromuscular function will be assessed by Barry-Albright Dystonia Scale score.
Gross Motor Function Measure | Baseline up to Month 24
  Neuromuscular function will be assessed by gross motor function measure.
Awake Oxygen Saturation Levels | Baseline up to Month 24
  Effect of EPI-743 on respiratory function will be measured by awake oxygen saturation levels.
Total Ventilator Days and Total Intensive Care Unit Days | Baseline up to Month 24
Number of Participants With Pneumonia Episodes and Tracheostomy | Baseline up to Month 24
Total Number of Mortalities, Medical Encounters, Hospitalizations, and Hospital Days | Baseline up to Month 24
Health-Related Quality of Life as Measured by NPMDS Section 4 Score | Baseline up to Month 24
Glutathione Cycle Biomarkers Level | Baseline up to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cohen, MD, Principal Investigator — Akron Children's Hospital
Locations (4):
- United States (4):
  - Gregory Enns, Stanford University, California
  - Akron Children's Hospital, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington